CLINICAL TRIAL: NCT02162524
Title: Effects of Images Following Long-term Aerobic Exercise on Brain Activation (E-Mechanic Ancillary II)
Brief Title: Effects of Images Following Long-term Aerobic Exercise on Brain Activation
Acronym: E-Mech Anc II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, John Apolzan, Postdoctoral Fellow, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 2013-045
Record Dates: First submitted 2013-09-17; First posted 2014-06-12 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: aerobic exercise; obesity; energy balance
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Exercise Control (No Intervention): Healthy Living Group
- Aerobic Exercise Group (Active Comparator): Persons are aerobically exercising.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — The exercise groups will be closely monitored during exercise sessions for six months in our exercise-training laboratory. The intensity will be 65% VO2peak and all exercise will occur on a treadmill. One exercise group will obtain 8 KKW (kcal/kg/week) over 3-4 sessions per week, which will result in each session lasting approximately 30 minutes. The other exercise group will obtain 20 KKW, performing 4-5 sessions per week for approximately 50-70 minutes per session. These groups are combined for this ancillary study.
  Other Names: 8KKW; 20KKW
  Arms: Aerobic Exercise Group

SUMMARY:
The primary purpose of this study is to quantify activation of regions of the brain associated with appetite and reward after viewing high sugar and high fat (HS/HF) images compared to control images following long-term aerobic exercise.

1. After long-term aerobic exercise compared to a no-exercise control group, viewing HS/HF food images vs. control images will result in higher activation of regions of the brain associate with appetite (hypothalamus).
2. After long-term aerobic exercise compared to a no-exercise control group consumption of a sucrose solution compared to an artificially sweetened solution and a tasteless solution, viewing HS/HF food images vs. control images will result in lower activation of regions of the brain associated with reward [amygdala, anterior cingulate cortex (ACC), Orbitalfrontal Cortex (OFC), and ventral tegmental area (VTA), striatum, insula] in overweight and obese men and women.

Exploratory Aims As exploratory aims, investigators will test a preliminary brain connectivity analysis.

DETAILED DESCRIPTION:
In this pilot study, investigators will use functional magnetic resonance imaging (fMRI) to determine the effects of high calorie visual food cues [i.e. images of foods that are high in both sugar and fat (HS/HF), such as ice cream] on activation of appetite and reward pathways in the brain following long-term (6 months) exercise. Obesity rates are high among US adults with 33.8% of adults having a BMI of 30 or greater (1). The prevailing belief is that homeostatic systems are in place to monitor energy homeostasis.

With aerobic physical activity, appetite is affected because a theoretically positive coupling between energy intake and expenditure is thought to occur (2, 3). During exercise days, short term studies have demonstrated that there are no differences in appetite except for a transient decrease 15 minutes post exercise after very hard exercise(4). Short term exercise does not result in appetitive differences (5-7). However in the medium term, there is a variable (mixed) response (5). Over the long-term it is thought a loose coupling exists between exercise and appetite response (5).

Our preliminary data strongly support a positive coupling between exercise and appetitive responses because in previous studies the amount of weight loss that is achieved following aerobic exercise is less than expected. Specifically, studies by Tim Church have previously found that hypertensive overweight postmenopausal women did not lose ~2.6 kg but instead 1.4 kg (8). This is a 46% difference between how much weight should be lost due to energy expended with exercise compared to the actual amount. Another study examined 4 months of moderate intensity aerobic exercise of 16KKW (9) and again about 2.7 kg of weight loss was expected but only 1.1 kg was achieved. This suggests a 59% difference. Both studies had very low dropout rates. Based on the results of the highest dose of exercise in these two studies, the discrepancy grows with an increase in exercise dose. The participants were instructed not to change eating habits and physical activity outside of the intervention and these were not significantly altered. These body weight responses mirror the majority of aerobic exercise intervention studies. King et al. performed a supervised aerobic exercise study (10). 58 persons completed 500 kcal/d of exercise induced energy expenditure for 5 d/wk over 12 weeks with a 28% dropout rate. Overall an average of just 3.2 kg of body weight was lost. Over 50% of persons failed to lose the expected amount and 15% of persons gained weight (11). Four out of ten studies in a review found exercise did not even result in a body weight difference between the exercise and control groups(12). This differential response in energy balance is thought to be driven by increased energy intake. Stubbs et al. performed a randomized crossover study with 3-7 day exercise treatments. The exercise treatments were no exercise, then medium exercise (~1.9 MJ/day) and lastly high exercise (~ 3.4MJ/day). Energy expenditure increased in the no exercise (9.2 MJ/day), medium exercise (11.0 MJ/day) and high exercise conditions (12.1 MJ/day), respectively. A statistically significant increase in energy intake with exercise was found (no exercise 8.9 MJ/day, medium exercise 9.2 MJ/day, and high exercise 10.0 MJ/d). Thus based on body weight and these energy intake data from Stubbs et al. investigators feel there is a biological drive to increase energy intake following exercise. Investigators seek to determine the neural mechanism of this appetitive response in the proposed grant.

Previously 2 aerobic exercise studies examining for the neuronal response to images have been performed. Ours are similar and will provide PBRC with pilot data for further investigations. Evero et al. previously found that reward pathway neuronal cues were reduced following aerobic exercise (13). Cornier et al. found that chronic exercise alters the neuronal response to food cues. However this study was confounded due to significant weight loss which as stated above does not generally happen with aerobic exercise trials. The results suggested the insula may be particularly important in exercise induced weight loss and weight loss maintenance (14). This study hopes to examine the neuronal responses to aerobic exercise without weight loss.

Obesity Women were shown food picture cues of high energy foods. The high energy foods produced significantly greater activation in the brain reward regions in obese compared to normal weight control women (15). Differences between groups included ACC, VTA, nucleus accumbens (NAc), amygdala, ventral pallidum (Vent Pall), Caudate, and Putamen (15). Postmeal, obese individuals, but not normal weight individuals, increase activation of the putamen (part of striatum) and amygdala suggesting these regions may play a role in overeating (16) which is why these regions are incorporated into the current study hypothesis. These cross-sectional studies are important as previously Murdaugh et. al (17) found that obese individuals that were not successful at short term weight loss or longer term weight loss maintenance had greater activation of reward pathway brain regions. While speculative, artificial sweeteners may reduce cravings by not activating reward pathways especially in obese persons. This grant will help provide pilot data to further elucidate this important question.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18-65 years old (inclusive)
* Weigh less than 350 lbs
* Body mass index (BMI) between 25-43 kg/m2
* Willing to fast for 10 hours prior to examination
* Right handed

Exclusion Criteria:

* Diagnosis (by self report) of diabetes
* Diagnosis (by self report) of neurological condition
* Current or past alcohol or drug abuse problem
* Smoking
* Have internal metal medical devices including cardiac pacemakers, aortic or cerebral aneurysm clips, artificial heart valves, ferromagnetic implants, shrapnel, wire sutures, joint replacements, bone or joint pins/rods/screws/clips, metal plates, metal fragments in your eye, or non-removable metal jewelry such as rings
* Unable or unwilling to complete the imaging procedures for the duration of the MRI scan due to claustrophobia or other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
fMRI | baseline and post (6 month intervention)
  fMRI will be performed using a General Electric Signa Excite HDxT 3.0T scanner (Milwaukee, WI) approximately 10 minutes post beverage ingestion. The field of view is 24-28 cm. The scanner is equipped with functional components from GE. Supplemental components include a projection system and eye imaging system from Avotec , Inc. An eight channel head coil will be utilized for all fMRI scans, and E-prime® software will be utilized for computerized experiment design, data collection, and analysis. Visual food and control cues will be presented in a mixed event block design with blocks of HS/HF and control images. Food cues consist of full-color pictures displaying foods within a category (HS/HF). One food item will be shown in each picture. Control cues consist of scrambled images that match the food cues in color intensity and frequency. Each block is 30s in length and 6 images are presented anywhere from 3-7seconds. Total task time will be ~30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — PBRC
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States